CLINICAL TRIAL: NCT04284540
Title: A Non-Randomized, Open-Label, Multi-Center Pilot Study Evaluating Hypofractionation Radiation Therapy in Head and Neck Squamous Cell Carcinoma
Brief Title: Hypofractionated Radiotherapy in Elderly Patients With Head & Neck Squamous Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Richard L. Bakst, Associate Professor, Radiation Oncology, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 19-0499
Record Dates: First submitted 2020-02-24; First posted 2020-02-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC)
Keywords: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma; Radiotherapy; Over 70 years of age; Elderly; shorter course of radiation treatment
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant Hypofractionated Radiation Treatment (Experimental): Short course radiation therapy for patients who have undergone surgery
  Interventions: Radiation: Adjuvant hypofractionation
- Definitive Hypofractionated Radiation Treatment (Experimental): Short course radiation therapy for patients who have not had surgery
  Interventions: Radiation: Definitive Hypofractionation

INTERVENTIONS:
Radiation: Adjuvant hypofractionation — 15 fractions of 2.7 Gy per fraction daily over 3 weeks for a total of 40.5 Gy to the post-operative bed and/or necks.
  Arms: Adjuvant Hypofractionated Radiation Treatment
Radiation: Definitive Hypofractionation — 15 fractions of 3 Gy per fraction daily over 3 weeks for a total of 45 Gy to regions of gross disease. Elective areas can be treated to 37.5 Gy in 15 fractions.
  Arms: Definitive Hypofractionated Radiation Treatment

SUMMARY:
The purpose of this research study is to investigate a shorter radiation treatment schedule for head and neck cancers in patients 70 years of age and older.

Standard radiation treatment for head and neck patients normally requires that the patient travel to the hospital daily for 6-7 weeks to receive radiation treatment 5 days per week. This long course of radiation can lead to significant side effects resulting in some people being unable to complete the course of treatment. If this happens, and there are gaps in the radiation treatment, this can lead to worse outcomes.

DETAILED DESCRIPTION:
This is a non-randomized pilot study examining the objective response rate and tolerability of short-course radiotherapy (RT) in elderly patients who are unfit for standard conventional fractionation treatment with head and neck squamous cell carcinoma (HNSCC). There will be two unrelated cohorts in this study: definitive RT and adjuvant RT. Patients will be assigned to the cohorts based on their surgical or non-surgical candidacy. The primary study measure is the locoregional control (LRC) rate of patients at 6 months post RT treated with short-course RT. Locoregional control at one year will be determined by radiographic (PET/CT) and clinical assessment of disease. For the definitive cohort, LRC will be defined as regression in size or disappearance of primary tumor and/or lymph nodes on imaging or clinical examination; and for the adjuvant cohort, LRC will be defined as absence of disease on imaging or no clinical evidence of disease.

To further investigate the treatment regimen, the study team will assess the safety of short-course RT and determine the incidence of serious complications, overall survival (OS), disease-free survival (DFS) within 1 year, and the change in quality of life (QoL) in these patients who are unfit for standard conventional fractionation treatment with head and neck squamous cell carcinoma (HNSCC) as secondary objectives. Secondary endpoints will include 1- year overall survival (OS), 1-year disease-free survival (DFS), and the total score of the Functional Assessment of Cancer Therapy-Head and Neck questionnaire (FACT-H&N). DFS will be defined from the completion of treatment until disease recurrence locally, regionally and/or distantly or until death from disease. OS will be defined from the RT to death or to last follow-up.

As a safety endpoint, the study team will calculate number and proportion of patients developing reportable AEs and SAEs according to relatedness to the treatment and stratified by severity.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 70 years.
* No previous RT or chemotherapy for HNSCC is allowed at time of study entry.
* Life expectancy > 12 weeks.
* Participants must have histologically or cytologically confirmed diagnosis of HNSCC: oral cavity, oropharynx, nasopharynx, hypopharynx, larynx, cervical nodes (unknown primary)
* All stages (according to National Comprehensive Cancer Network 8th edition for head and neck cancers), except stage IVC5
* Non-concurrent chemotherapy
* First line treatment
* Anyone eligible for definitive or adjuvant based RT therapy
* Adjuvant therapy when histopathological factors (advanced T category, nodal disease, lymphovascular or perineural invasion, high-grade, or positive margins)
* Anyone being treated with curative intent
* Unfit as determined by the treating physician and ECOG performance 1, 2, or 3 (Appendix 2).
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria

* Patients < 70
* Metastatic disease outside of the head and neck
* Pregnancy
* Previous or current malignancies at other sites, with the exception of adequately treated in situ carcinoma of the cervix, basal or squamous cell carcinoma of the skin, thyroid cancer, or other cancer curatively treated by surgery and with no current evidence of disease for at least 5 years.
* Prior RT of head and neck area
* Concurrent chemotherapy or immunotherapy or hormonotherapy
* Any comorbid connective tissue disorder which could aggravate RT associated toxicities (e.g. Scleroderma)
* In cases where patients cannot consent on their own due to underlying dementia, we can consent the patient's healthcare proxy

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with Locoregional Control (LRC) | 6 months
  For the adjuvant cohort: LRC will be defined as absence of disease on imaging or no clinical evidence of disease. For the definitive cohort: LRC will be defined as regression in size or disappearance of primary tumor and/or lymph nodes on imaging or clinical examination.

SECONDARY OUTCOMES:
Overall Survival (OS) rate | 1 year
  1 year overall survival of patients as defined by completion of treatment until death at 1 year.
Disease Free Survival (DFS) rate | 1 year
  1 year disease free survival of patients as defined by completion of treatment until disease recurrence locally, regionally and/or distantly or until the time of death due to disease assessed via PET scan and physical exam.
University of Washington Quality of Life Questionnaire (UW-QOL) | Up to 3 years
  University of Washington Quality of Life Questionnaire (UW-QOL) full scale from 0 to 100, with higher score indicating poorer health outcomes.
FACT-H&N questionnaire | Up to 1 year
  Foundation for the Accreditation of Cellular Therapy-Head and Neck (FACT-H&N) questionnaire, 38-item instrument. Full scale from 0 to 144, with higher score indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Richard L. Bakst, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - Mount Sinai Downtown Union Square, New York, New York
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No
All of the individual participant data collected during the trial, after deidentification.